CLINICAL TRIAL: NCT04618432
Title: Collection of Clinical Data and Specimens for Research on Head and Neck and Communication Disorders
Status: Terminated | Type: Observational
Why Stopped: PI moved institutes in NIH, and this protocol was redundant with an existing clinical protocol within the new institute.
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000077; 000077-DC
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Carcinoma
Keywords: Carcinoma; Hearing; Balance; Neoplasm; Natural History
MeSH Terms: conditions — Carcinoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients at risk, suspected of having, have a history of, or currently have a diagnosed head and neck or communication disorder.

SUMMARY:
Study Description:

It may be in the interest of the NIDCD Clinical Research Program (CRP) to collect clinical data or specimens generated in the diagnosis and treatment of head and neck or communication disorders and to evaluate patients to determine candidacy for intramural clinical studies. This protocol will provide the administrative vehicle to enable the evaluation and provision of clinical care for patients with head and neck and communication disorders by the NIDCD CRP, Clinical Center, and consult services. No investigational therapies will be administered in this

study.

Objectives and Endpoints:

(Summation)To collect clinical data or specimens generated in the diagnosis and treatment of head and neck or communication disorders

(Summation)To evaluate patients to determine candidacy for intramural clinical studies

Study Population:

Patients at risk, suspected of having, have a history of, or currently have a diagnosed head and neck or communication disorder referred to NIDCD Clinical Investigators by the Intramural Consult Service or community providers

Description of Sites:

NIH Clinical Center

Study Duration:

10 years

DETAILED DESCRIPTION:
Study Description:

It may be in the interest of the NIDCD Clinical Research Program (CRP) to collect clinical data or specimens generated in the diagnosis and treatment of head and neck or communication disorders and to evaluate patients to determine candidacy for intramural clinical studies. This protocol will provide the administrative vehicle to enable the evaluation and provision of clinical care for patients with head and neck and communication disorders by the NIDCD CRP, Clinical Center, and consult services. No investigational therapies will be administered in this

study.

Objectives and Endpoints:

(Summation)To collect clinical data or specimens generated in the diagnosis and treatment of head and neck or communication disorders

(Summation)To evaluate patients to determine candidacy for intramural clinical studies

Study Population:

Patients at risk, suspected of having, have a history of, or currently have a diagnosed head and neck or communication disorder referred to NIDCD Clinical Investigators by the Intramural Consult Service or community providers

Description of Sites:

NIH Clinical Center

Study Duration:

10 years

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must be age 2 years or older if procedures or treatment are required.
* Patients at risk, suspected of having, have a history of, or currently have a diagnosed head and neck or communication disorder.
* An NIDCD clinical investigator and PI determines it is in the interest of the patient/individual and NIDCD CRP for the subject to undergo consult, treatment or follow-up at the NIDCD/NIH
* Patient or their Legally Authorized Representative is able to provide informed consent.

EXCLUSION CRITERIA:

* Candidates who do not meet the inclusion criteria.
* Candidates who in the opinion of the PI and clinical team have medical or unstable conditions for which NIDCD and CC consultative services are unable to provide or support optimal care

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at risk, suspected of having, have a history of, or currently have a diagnosed head and neck or communication disorder referred to NIDCD Clinical Investigators by the Intramural Consult Service or community providers
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Evaluation for clinical studies | ongoing
  To evaluate patients to determine candidacy for intramural clinical studies
Clinical data collection | ongoing
  To collect clinical data or specimens generated in the diagnosis and treatment of head and neck or communication disorders

CONTACTS AND LOCATIONS:
Overall Officials: Clint T Allen, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000077-DC.html